CLINICAL TRIAL: NCT01621230
Title: A Randomized Double-blinded Trial of the Effects of Bupivacaine Induced Motor Blockade on the Second Stage of Labor
Brief Title: Effects of Bupivacaine Induced Motor Blockade During the Second Stage of Labor
Acronym: BUP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Margaret Craig, Primary Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU 042011-045
Record Dates: First submitted 2012-02-06; First posted 2012-06-18 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Pregnancy
Keywords: Bupivacaine; Fentanyl; Epidural; Second Stage of Labor; Randomized Controlled Trial
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: double-blinded 2 arm
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural fentanyl (Active Comparator): A continuous epidural infusion of fentanyl 10 mcg/cc at a basal infusion rate of 10 ml/hr with a patient-controlled epidural analgesia (PCEA) demand dose of 5 mL/hr for pain. Meperidine 25 mg intravenously every 1 hour for breakthrough pain as needed.
  Interventions: Drug: Epidural fentanyl
- Epidural bupivacaine plus fentanyl (Placebo Comparator): A continuous epidural infusion of bupivacaine plus fentanyl during the second stage (i.e. 10 cm dilation) of labor. Epidural infusion are 10 ml/hr basal infusion plus 5 ml/hr demand dose via patient-controlled epidural analgesia (PCEA). Meperidine 25 mg intravenously every 1 hour for breakthrough pain as needed .
  Interventions: Drug: Epidural Bupivacaine plus fentanyl

INTERVENTIONS:
Drug: Epidural Bupivacaine plus fentanyl — The subjects will receive 0.125% bupivacaine with fentanyl 2 mcg/mL at a rate of 10 mL/hr.
  Other Names: Epidural continous infusion of bupivacaine and fentanyl
  Arms: Epidural bupivacaine plus fentanyl
Drug: Epidural fentanyl — The subjects will receive epidural fentanyl 10 mcg/mL with the rate of 10mL/hr.
  Other Names: Epidural continous infusion of fentanyl
  Arms: Epidural fentanyl

SUMMARY:
The aim of this study is to measure the effects of bupivacaine administered via epidural catheters on indices of motor blockade ascertained during the second stage of labor. This is a randomized, double-blind, controlled trial designed to address the primary research question: Does bupivacaine lengthen the second stage of labor? The secondary research question is: Is there other evidence of motor blockade attributable to bupivacaine during the second stage of labor?

The investigators know from prior studies that the length of the second stage in nulliparous women delivered at Parkland Hospital without epidural analgesia is 28 minutes. The investigators hypothesize in this now proposed study that epidural analgesia with bupivacaine will significantly increase this baseline from 28 minutes to 37 minutes or more (a 33% increase) thus implicating motor blockade. Baseline data for the Bromage and Breen scores during the second stage as well as the uterine contractility data are not available as these indices of motor blockade have not here-to-fore been studied in this context.

Currently at Parkland Hospital, 82% of nulliparous women undergoing induction of labor at term receive continuous epidural infusions with bupivacaine during the first and second stages of labor. Such women will be identified when admitted for scheduled inductions at Parkland. After informed consent is obtained standard management of labor induction will be provided. Those consented women reaching 8 cm cervical dilation will be randomized. Group I will receive bupivacaine plus fentanyl via epidural catheter during the second stage (i.e. 10 cm dilation) and Group II will receive only fentanyl infusion via epidural catheter (see study procedure below). Both the patient and the caregiver will be blinded as to whether the patient is in the bupivacaine plus fentanyl arm or the fentanyl only arm. To detect a 33% increase (from 28 minutes to 37 minutes) in the primary outcome the investigators need a total of 310 women enrolled in the study (or 155 per arm). Assuming a 30% consent rate and given that approximately 1000 women meet the inclusion criteria each year at Parkland, the investigators project that this study could be completed in 12 months.

DETAILED DESCRIPTION:
Nulliparous women scheduled for labor inductions on Monday through Friday and who have consented to this study will be randomized to one of two arms: bupivacaine plus fentanyl epidural analgesia throughout labor and delivery (including the second stage) or epidural bupivacaine plus fentanyl until 8 cm cervical dilation and only fentanyl thereafter. From activation of epidural analgesia to 8 cm cervical dilation the prevailing standard epidural technique in use at Parkland Hospital will be used. Briefly, 19-ga multi-orifice epidural catheter is placed using 17-ga 3 ½cm Tuohy needle into the L3-L4 lumbar interspace. Lactated Ringers solution, 500-1000mL will be infused during placement of the epidural catheter to mitigate hypotension. A test dose using 1.5% lidocaine with 1:200,000 epinephrine, 3mL, will be given via the epidural catheter. If the test dose is negative, then an initial bolus of 0.25% bupivacaine, 4-8mL, with fentanyl 100mcg is given via the catheter. After securing the epidural catheter the patient will be placed in the supine position and the anesthetic sensory level measured with the desired level of T6-T8. Once a T6-T8 sensory block is secured the epidural infusion using 0.125% bupivacaine with 2mcg/mL fentanyl at 10mL/hr will be started.

At any time during epidural infusion the epidural catheter may be replaced at the discretion of the anesthesia provider for inadequate analgesia. Ephedrine or phenylephrine will be given intravenously for maternal hypotension defined as systolic blood pressure ≤ 90 mmHg or a decrease of 20% systolic blood pressure from patient's baseline.

Randomization will occur when the woman reaches 8 cm cervical dilation. Envelopes containing cassettes will be sequentially randomized by Dr. McIntire and given to the attending obstetrical anesthesiologist containing one of two medications. Group I will receive a 100mL epidural cassette of 0.125% bupivacaine with fentanyl 2mcg/mL to be infused at 10mL/hr. Group II will receive a 100mL cassette of fentanyl 10mcg/mL (to be infused at 10mL/hr. Both groups will have the same rate of epidural infusion such that the patient, nurse, obstetrician, and anesthesia providers will be blinded to the randomized treatment group. The Parkland Investigational Drug Service (IDS) will provide the study drugs.

The patient may request a 5mL bolus from the epidural infusion every 30 minutes if pain relief is inadequate. The obstetrician can also give patients in either study group 25mg of intravenous meperidine every hour for up to two doses if pain relief is unsatisfactory. The study regimen will continue until spontaneous delivery of the infant or until which time operative vaginal delivery or cesarean delivery is planned. At this point the study will be over and routine anesthesia care resumed.

The standard of care for management of labor induction at Parkland requires continuous electronic fetal heart rate monitoring (EFM) as well as uterine contraction monitoring. The standard is to apply EFM internal transducers when the membranes are ruptured. Standard fetal monitors equipped with laptop computers will be used to electronically store the fetal heart rate and uterine contraction data during this study. This will permit qualification of uterine contractility during the second stage of labor. The Bromage and Breen scores for motor blockade will be assessed at complete cervical dilation and at 30, 60, and 90 minutes thereafter. The scoring system is as follows:

Score Criteria

1. Unable to move feet or knees (complete block)
2. Able to move feet only
3. Just able to move knees
4. Detectable weakness of hip flexion while supine
5. No weakness of hip flexion
6. Able to perform partial knee bend

Visual analog pain (VAS) scores for the adequacy of epidural analgesia from 1-10 will also be assessed at each time point used for the Bromage and Breen scores.

Data collection will include maternal demographic characteristics as well as antepartum and intrapartum obstetrical features. Condition of the infant at birth based on Apgar scores and umbilical artery blood pH, as well as neonatal outcomes will be ascertained.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women at 37 weeks gestation or greater.
* Scheduled for induction of labor for any indication, to include hypertensive disorders, diabetes, decreased fetal motion, or prolonged pregnancy.
* Single without known malformations.
* Maternal age > or equal to 16 years.
* ASA classification 1 or 2.

Exclusion Criteria:

* Women who refuse epidural analgesia.
* Women with contraindications to epidural analgesia, i.e., severe thrombocytopenia.
* Any renal disease with serum creatinine > 1.0 mg/dL.
* Allergy to bupivacaine or fentanyl.
* Known liver disease such as hepatitis.
* Known contraindications to internal electronic fetal monitoring i.e., active herpes, maternal HIV seropositivity.

Ages: 16 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 481 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Leveno, MD, Study Chair — University of Texas Southwestern Medical Center; Lisa Moseley, Study Director — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health and Hospital System, Dallas, Texas, United States

REFERENCES:
- [Result] Craig MG, Grant EN, Tao W, McIntire DD, Leveno KJ. A randomized control trial of bupivacaine and fentanyl versus fentanyl-only for epidural analgesia during the second stage of labor. Anesthesiology. 2015 Jan;122(1):172-7. doi: 10.1097/ALN.0000000000000454. PMID 25254902

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1,013 women met the study inclusion criteria between September 7, 2009 and July 16, 2012 at Parkland Hospital. A total of 481 women were consented to participate in the study, and 310 women were randomized to receive the allotted study drug. The remaining women delivered without receiving an epidural.
Pre-assignment Details: 171 women delivered prior to randomization at 8 cm cervical dilation.
Groups:
- Bupivacaine Plus Fentanyl: Group I received bupivacaine plus fentanyl via epidural catheter during the second stage (i.e. 10 cm dilation) of labor via continuous epidural infusion of 10 cc/hr basal infusion plus 5 cc/hr demand dose via patient-controlled epidural analgesia (PCEA). Group I was allowed to receive meperidine 25 mg iv q1 hour for breakthrough pain.
- Fentanyl Only: Group II received a continuous infusion of fentanyl 10 mcg/cc at a basal infusion rate of 10 cc/hr with a patient-controlled epidural analgesia (PCEA) demand dose of 5 cc/hr for pain. Group II (like Group I) received meperidine 25 mg iv for breakthrough pain as needed.
Period: Overall Study
Arm/Group | Bupivacaine Plus Fentanyl | Fentanyl Only
Started | 154 | 156
Completed | 154 | 156
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Plus Fentanyl | Fentanyl Only | Total
Number analyzed (Participants) | 154 | 156 | 310
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 154 | 156 | 310
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.6 (5.4) | 22.9 (5.0) | 22.7 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 156 | 310
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 154 | 156 | 310

OUTCOME MEASURES:

1. Primary Outcome: The Duration of the Second Stage of Labor
Description: The length of the second stage of labor (measured as minutes a parturient spends in Stage II) in nulliparous women received a epidural bupivacaine plus fentanyl or fentanyl alone.
Time Frame: Duration of second stage of labor approximately 30 minutes to 150 minutes
Measure: Median (Full Range); unit: minutes
Groups:
- Group I (Bupivacaine): Group I received bupivacaine plus fentanyl via epidural catheter during the second stage (i.e. 10 cm dilation) of labor via continuous epidural infusion of 10 cc/hr basal infusion plus 5 cc/hr demand dose via patient-controlled epidural analgesia (PCEA). Group I was allowed to receive meperidine 25 mg iv q1 hour for breakthrough pain.
- Group II (No Bupivacaine): Group II received a continuous infusion of fentanyl 10 mcg/cc at a basal infusion rate of 10 cc/hr with a patient-controlled epidural analgesia (PCEA) demand dose of 5 cc/hr for pain. Group II (like Group I) received meperidine 25 mg iv for breakthrough pain as needed.
Arm/Group | Group I (Bupivacaine) | Group II (No Bupivacaine)
Number analyzed (Participants) | 154 | 156
minutes | 75 [41 to 128] | 73 [42 to 120]
Statistical Analysis 1: Comparison: Group I (Bupivacaine) vs Group II (No Bupivacaine); Test type: Other — The median (first and third quartile) lengths of the second stage of labor were estimated at 28min (15, 58) in women without epidural analgesia. Assuming a one-third increase in the length of the second stage to 37min due to epidural bupivacaine, a sample size of 155 per arm (310 total) was required for 80% power to detect such a difference using a two-sided Wilcoxon rank sum test; p = 0.17, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Local Anesthetic Motor Blockade Indices During Stage II of Labor
Description: Motor blockade will be estimated using Bromage and Breen scores (measured on a 6-point standardized scale, 1= Unable to more feet, 6= Able to perform partial knee bend) that estimate motor blockade. This scoring system is based upon the laboring womans' ability to move her lower extremities.
Time Frame: Duration of second stage of labor approximately 30 minutes to 150 minutes
Population: PI for this study is deceased and the relevant data have been destroyed. The underlying data are not available for accurately reporting the information in this Outcome Measure
Groups:
- Epidural Bupivacaine Plus Fentanyl (Bupivacaine): A continuous epidural infusion of bupivacaine plus fentanyl during the second stage (i.e. 10 cm dilation) of labor. Epidural infusion are 10 ml/hr basal infusion plus 5 ml/hr demand dose via patient-controlled epidural analgesia (PCEA). Meperidine 25 mg intravenously every 1 hour for breakthrough pain as needed .
  Epidural Bupivacaine plus fentanyl: The subjects will receive 0.125% bupivacaine with fentanyl 2 mcg/mL at a rate of 10 mL/hr.
Arm/Group | Epidural Bupivacaine Plus Fentanyl (Bupivacaine)
Number analyzed (Participants) | 0

3. Secondary Outcome: Mode of Delivery in Women Randomized to Bupivacaine vs. No Bupivacaine During the Second Stage of Labor
Time Frame: At the time of Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Fentanyl | Epidural Bupivacaine Plus Fentanyl (Bupivacaine)
Number analyzed (Participants) | 156 | 154
Participants
  Spontaneous | 126 | 112
  Forceps-assisted | 12 | 19
  Cesarean | 18 | 23

4. Secondary Outcome: Number of Participants Whose Newborns Received an APGAR Score of <=3 at 1 Min
Description: Number of participants whose newborns received an APGAR score of <=3 at 1 min. A lower APGAR score represents poor health or a worsening in the Outcome,
Time Frame: At the time of Delivery, up to 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Fentanyl | Epidural Bupivacaine Plus Fentanyl (Bupivacaine)
Number analyzed (Participants) | 156 | 154
Participants | 14 | 11
Statistical Analysis 1: Comparison: Epidural Fentanyl vs Epidural Bupivacaine Plus Fentanyl (Bupivacaine); Test type: Other; p = .55, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants Whose Newborns Received an APGAR Score of <=3 at 5 Min
Description: Number of participants whose newborns received an APGAR score of <=3 at 5 minutes. A lower APGAR score represents poor health or a worsening in the Outcome
Time Frame: At the time of Delivery, up to 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Fentanyl | Epidural Bupivacaine Plus Fentanyl (Bupivacaine)
Number analyzed (Participants) | 156 | 154
Participants | 2 | 1
Statistical Analysis 1: Comparison: Epidural Fentanyl vs Epidural Bupivacaine Plus Fentanyl (Bupivacaine); Test type: Other; p = .57, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during study period start from beginning of the labor until the discharge from the hospital which was for the duration of labor (this time period varied for each participant), and then for 48 hours post-delivery (the normal timeframe when a woman is discharged from the hospital post-delivery).
Groups:
- Bupivacaine Plus Fentanyl: A continuous epidural infusion of bupivacaine plus fentanyl during the second stage (i.e. 10 cm dilation) of labor at a rate of 10 ml/hr basal infusion plus 5 ml/hr demand dose via patient-controlled epidural analgesia (PCEA). Subjects were allowed to receive intravenous meperidine 25 mg for breakthrough pain as needed.
- Fentanyl Alone: A continuous infusion of fentanyl 10 mcg/mL at a basal infusion rate of 10 ml/hr. and a demand dose of 5 ml/hr for pain. Subjects received intravenous meperidine 25 mg for breakthrough pain as needed.
Arm/Group | Bupivacaine Plus Fentanyl | Fentanyl Alone
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/156
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/156
Other Adverse Events (participants affected / at risk) | 0/154 | 0/156

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes